CLINICAL TRIAL: NCT04224948
Title: The PET-RPS Study: Utility of PET for Assessment of Response to Preoperative Chemotherapy in Primary Retroperitoneal Sarcoma (RPS)
Brief Title: The PET- Retroperitoneal Sarcoma Study
Acronym: PET-RPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 19-5429
Record Dates: First submitted 2019-07-04; First posted 2020-01-13 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Retroperitoneal Sarcoma
Keywords: Retroperitoneal Sarcoma; Retroperitoneal; Sarcoma; Neoadjuvant Chemotherapy; preoperative Chemotherapy
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- PET-MR arm (Experimental): Every eligible patient will be scanned by PET-MR at baseline and following 1 cycle of chemotherapy. PET-CT at baseline will also be obtained as it is the current standard of care and will be used to determine trial eligibility (no evidence metastasis at baseline).
  Interventions: Device: PET MRI scan

INTERVENTIONS:
Device: PET MRI scan — Standard of care includes a baseline PET-CT and conventional CT after 2 cycles of neoadjuvant chemotherapy, and after 5-6 cycles, of neoadjuvant chemotherapy, as per current practice/ standard of care.
  Patients that enroll in the trial will receive two additional PET MRI scans- one at baseline and one after 1 cycle of chemotherapy

SUMMARY:
Retroperitoneal sarcoma(RPS) is a rare cancer that is difficult to cure as it typically presents as a very large abdominal mass, and complete removal with clear margins is challenging . This study will focus on improving the outcomes of surgery by treating RPS before surgery, to make resection more effective. The role of chemotherapy as a preoperative treatment for RPS is highly controversial. Response to chemotherapy is unpredictable and if the patient's tumour progresses instead of responding, the window of opportunity for resection will be lost. Conventional cross sectional imaging (CT scan) is inadequate to measure response to chemotherapy until 5-6 cycles have been given, possibly with no improvement. Thus it is critical to develop an earlier and reliable way to assess response. Functional imaging by PET scan is used in other tumour types to identify early response to treatment. PET imaging may provide a more meaningful assessment of RPS response to systemic therapy much earlier in the course of treatment than conventional imaging, allowing timely modification of the treatment plan. This study will define the role of PET imaging in evaluating early response to systemic therapy in high grade RPS, improving patient treatment.

DETAILED DESCRIPTION:
Soft tissue sarcomas (STS) are derived from mesenchymal cells, and can arise at any site. Retroperitoneal sarcomas (RPS) account for ~15% of STS, and patients have much worse survival outcomes than for extremity STS. Local (abdominal) recurrence of RPS is very common, due to the challenges of obtaining complete resection of these large masses that abut critical central compartment structures, such as the inferior vena cava and aorta. There is currently intense interest in using preoperative therapy to downsize/cytoreduce RPS and hopefully improve oncologic outcomes. Studies have shown that preoperative radiation does not cytoreduce these tumours. In this study, the potential of systemic therapy for cytoreduction will be examined.

The standard systemic therapy regimen for treatment of patients with STS remains Adriamycin/Ifosphamide, although side effects can be tolerated only by relatively young and fit patients. The use of this regimen preoperatively for extremity STS results in average response rates of about 30-40%, as judged by histologic assessment of the resected specimen. The international experience with preoperative chemotherapy for RPS is very limited, and there are no published reports.

Functional imaging may provide a more meaningful assessment of tumour response to systemic therapy. PET-MR is a newer modality that may hold promise in assessing solid tumour response and its potential utility is currently of rapidly growing interest. Conventional MRI can offer a more detailed assessment of tumour relationships to adjacent structures than can CT, particularly in STS. Integration of PET with MR has the potential to provide information about metabolic tumour volume (MTV) and to help guide surgical planning.There are no data available on the utility of PET-MR in evaluating tumour response to chemotherapy in STS.

At present, the role of chemotherapy as a preoperative treatment for retroperitoneal sarcoma (RPS) is undefined and controversial. The sarcoma group at Princess Margaret Cancer Centre (PMCC) has had some experience with this treatment paradigm, but like most sarcoma groups in Ontario, and Canada, has reserved preoperative chemotherapy for frankly unresectable and borderline resectable tumours for which downsizing would potentially render resection more feasible. At present, CT-scan imaging is performed after 2 cycles of chemotherapy, and if there is no frank progression of the cancer, chemotherapy is continued for another 3-4 cycles. By that point the tumour is smaller on CT scan in about 30% of patients. There are 2 main problems with this approach: 1)70% of the patients may have undergone 5-6 cycles of chemotherapy with no apparent benefit; and 2) there may be a metabolic response and associated benefit without a change in tumour size. The ability to reliably assess tumour response earlier on (i.e. after 1 cycle) would significantly influence the care of these patients as ineffective chemotherapy could be terminated after 1 cycle and the regimen could be modified, or surgery could happen right away before the window of resectability is lost.

ELIGIBILITY:
Inclusion Criteria:

* Tumour-related criteria
* Primary soft tissue sarcoma of retroperitoneal space or infra-peritoneal spaces of pelvis
* Sarcoma not originated from bone structure, abdominal or gynecological viscera
* Unifocal tumour (not multifocal disease)
* Absence of extension through the sciatic notch or across the diaphragm
* Histologically-proven RPS (local pathologist/ imaging-guided or surgical biopsy), only including the following histological sub-types:
* High grade Leiomyosarcoma
* High grade Dedifferentiated Liposarcoma
* Tumour not previously treated (no previous surgery -excluding diagnosis biopsy-, radiotherapy or systemic therapy)
* Tumour both operable and suitable for chemotherapy (This will be based on pretreatment CT scan/MRI and multidisciplinary consultation with surgeon medical oncologist and radiologist (anticipated macroscopically complete resection, R0/R1resection)
* Patients for whom surgery is expected to be R2 on the CT-scan before randomization are not eligible
* Patients must have American Society of Anesthesiologist (ASA) score ≤ 2 (see Appendix G)
* The criteria for non-resectability are:
* (i) involvement of superior mesenteric artery
* (ii) involvement of aorta
* (iii) involvement of bone
* distant metastatic disease
* Patient must have radiologically measurable disease (RECIST 1.1)

Patient-related criteria

* ≥ 18 years' old
* WHO performance status ≤ 2 (see Appendix C)
* Absence of history of bowel obstruction or mesenteric ischemia or severe chronic inflammatory bowel disease
* Normal renal function:
* Calculated creatinine clearance within normal value Functional contra-lateral kidney to the side involved by the RPS as assessed by intravenous pyelogram (done during the baseline CT-scan) or differential renal isotope scan
* Normal bone marrow and hepatic function:
* White Blood cells ≥ 2.5 x10 9 cells/L
* Platelets ≥ 80 x10 9 cells/L
* Total bilirubin < 1.5 time the institutional upper limit normal of value (ULN)
* Adequate cardiac function: less or equal to NYHA II
* Normal 12 lead ECG (without clinically significant abnormalities)
* No co-existing malignancy within the last 5 years except for adequately treated basal cell carcinoma of the skin or carcinoma in situ of the cervix
* No prior abdominal or pelvic irradiation for other prior malignancy or other disease
* Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule
* Excluding patients who presented after incomplete resection and underwent immediate completion surgery.

Exclusion Criteria:

* Age< 18 years
* Recurrent tumour
* Benign retroperitoneal tumours
* Presence of second active cancer
* Serious psychiatric disease that precludes informed consent or limits compliance
* impossible to ensure adequate follow up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-01-03 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Correlation of PET imaging with histologic response following preoperative chemotherapy. | 3 years
  Pathology of RPS specimens, resected following standard ifosfamide/doxorubicin chemotherapy every 3 weeks for 5-6 cycles, will be compared with PET response (FDG uptake) after cycle 1 of chemotherapy.

SECONDARY OUTCOMES:
Correlation of CT imaging with histologic response, and comparing prognostic accuracy of PET-MR vs.CT imaging for histologic response, recurrence status, and survival. | 3 years
  Pathology of resected RPS specimens, resected following standard ifosfamide/doxorubicin chemotherapy every 3 weeks for 5-6 cycles, will be compared with CT response after 2 and 5/6 cycles of preoperative chemotherapy. PET imaging and CT imaging will be compared as prognosticators of histological response, recurrence and survival.

CONTACTS AND LOCATIONS:
Overall Officials: Carol Swallow, MD, PhD, Principal Investigator — Sinai Health System
Locations (1):
- University Health Network and The Sinai Health System, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No